CLINICAL TRIAL: NCT00868049
Title: Study of Stomatognathic System,Chewing and Deglutition Functions in the Obese Subjects
Brief Title: Study of Stomatognathic System of the Obese Subjects
Acronym: SSSCDFO
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Adriana Bueno de Figueiredo/ Master Student, Clinic Hospital of Medical School of University of Sao Paulo
Other Study IDs: ADRIANABF1
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: chewing; deglutition; orofacial motricity; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Obese subjects
- 2: Normal-weight subjects

SUMMARY:
The aim is to identify differences in the stomatognathic system, mastication and deglutition functions between obese and normal weight subjects.

DETAILED DESCRIPTION:
The aim of this study was to identify differences in the stomatognathic system between obese and normal weight subjects. The habitual chewing of a French bread and deglutition of solids and liquid was evaluated five times in obese subjects and controls. The tonus of the lips, tongue, cheeks, masseter and temporal muscles were evaluated by clinical observation and palpation and defined as either normal or reduced. Twenty obese patients (body mass index (BMI) > 30kg/m2) and twenty volunteers of normal weight (BMI 18.5-24.9 Kg/m2) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults male and female
* healthy dentate
* body mass index (BMI) higher than 30 Kg/m2 for the obesity group and (BMI) lower than 25/m2 for the normal weight group.

Exclusion Criteria:

* face deformity
* alterations in morphology of lips and tongue
* without teeth or with lack of one tooth (excluding third molars)
* Malocclusion Angle's Class II and III
* pain during chewing
* pathology of the temporomandibular joint
* neurological pathology

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: twenty obese patients (6 Male /14 Female, mean age 32.2 ± 9.9, mean BMI 43,3 ± 9.6 Kg/m2) and twenty lean volunteer (4 Male / 16 Female mean age 30.7 ±6.7, mean BMI 22.3 ± 1.9 Kg/m2)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana B Figueiredo, MS, Principal Investigator — Clinic Hospital of Medical School of University of São Paulo
Locations (1):
- Medical School of University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Valera FC, Trawitzki LV, Anselmo-Lima WT. Myofunctional evaluation after surgery for tonsils hypertrophy and its correlation to breathing pattern: a 2-year-follow up. Int J Pediatr Otorhinolaryngol. 2006 Feb;70(2):221-5. doi: 10.1016/j.ijporl.2005.06.005. Epub 2005 Jul 21. PMID 16039726